CLINICAL TRIAL: NCT02083120
Title: Efficacy and Physiology of Nasal High Flow Therapy (AIRVO2™, Fisher&Paykel) in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Chronic Hypercapnic Respiratory Failure
Brief Title: Efficacy and Physiology of Nasal High Flow Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Georg Nilius, Head of pneumologic department of Helios Klinik Hagen, Helios Klinik Ambrock
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AIRVOhome
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: high flow; COPD; AIRVO
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nasal High Flow and Oxygen (Experimental): overnight nasal High Flow (NHF) therapy+ individually titrated supplemental oxygen (2-6 L/min),total 35 L/min, 4 weeks at home
  Interventions: Device: NHF therapy; Other: Long term Oxygen Therapy (LOT)
- Long term Oxygen Therapy (LOT) (Active Comparator): individually titrated supplemental oxygen (2-6 L/min), 4 weeks at home
  Interventions: Other: Long term Oxygen Therapy (LOT)

INTERVENTIONS:
Device: NHF therapy — AIRVO 2 device therapy is either a humidifier with integrated flow generator that delivers warmed and humidified respiratory gases to spontaneously breathing patients through a variety of patient interfaces. Flow rates up to 60 L/min are available to the user, depending on the patient interface and mode of operation.In this study, flow rates of 20 L/min and 35 L/min will be compared.
  Other Names: AIRVO 2; myAIRVO 2; PT101; PT100
  Arms: nasal High Flow and Oxygen
Other: Long term Oxygen Therapy (LOT) — Oxygen will individually be added to NHF in order to achieve stable oxygen saturation by pulse oximetry (SpO2) values of 88% to 92%.
  Other Names: supplemental oxygen

SUMMARY:
The effects of a nasal high-flow (NHF) therapy in patients with chronic obstructive hypercapnic respiratory failure are still not sufficiently known yet.

The aim of this study is a step-by-step generation of physiological data about gas exchange and respiration under high flow therapy using a nasal cannula with an AIRVO 2 device to provide NHF, leading to an analysis of the effects of high flow on PCO2 levels, exercise capacity, quality of life and gas exchange in a long term home treatment compared to a standard low flow long term oxygen therapy (LOT).

Hypothesis: NHF and LOT therapy show differences in measured mean overnight transcutaneous carbon dioxide partial pressure (PCO2) after four weeks of treatment.

DETAILED DESCRIPTION:
Stage 1: Respiratory Physiology. Aim of this Stage is to investigate the effects of nasal High Flow (NHF) therapy in patients in progressed stages of COPD, by measuring physiologic parameters like tidal volume, breathing frequency and expiratory PCO2 concentration.

Stage 2: Efficacy of short term NHF. Aim of this Stage is to evaluate the efficacy of two flow rates (20 L/min and 35 L/min) regarding alveolar ventilation in overnight therapy. For this reason, patients will have two PSG sleep studies during their hospital stay, under 20 L/min and 35 L/min NHF therapy in randomized order.

Stage 3: Home Care monitoring. Aim of this Stage is to compare long term influences of NHF and LOT on PCO2 levels randomised crossover, 4 weeks each treatment.

Stage 4: Long Term Home Care monitoring . Aim of this stage is the long term follow up (12 month) of patients to examine the compliance of a sufficient NHF therapy. Patients will retain the NHF therapy if they are responders (PCO2 improvement in stage 3 of at least 2 mmHG with NHF versus LOT) and willing and able to use NHF and a patient log.

All patients will be monitored for the next 12 month. After 6 month there will be a control phone call.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80
* Male and female
* COPD patients with chronic respiratory insufficiency (pH >7.35 and PCO2 > 50mmHg)
* Stable respiratory situation

Exclusion Criteria:

* Decompensated heart, liver or kidney failure.
* Pregnancy or nursing period
* Participation in another clinical trial within the last 4 weeks
* Drug abuse
* Incapable of giving consent
* Known obstructive sleep apnea syndrome (OSA) (AHI>10)
* noninvasive ventilation (NIV) therapy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04; Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
mean overnight transcutaneous PCO2 | baseline
  In two baseline measurements the aim is to evaluate the efficacy of two flow rates (20 L/min and 35 L/min) regarding alveolar ventilation in overnight therapy. For this reason, patients will have two polysomnographic sleep studies (PSG) during their hospital stay, under 20 L/min and 35 L/min NHF therapy in randomized order.
  Primary objective is the mean overnight transcutaneous PCO2 value, absolute as well as time spent >50 mmHg.
mean overnight transcutaneous PCO2 | after 4 weeks
  In home care monitoring is the aim to compare long term influences of NHF and LOT on PCO2 levels. Primary objective is the mean overnight transcutaneous PCO2 level measured after 4 weeks of each treatment phase.
mean overnight transcutaneous PCO2 | after 12 month
  All patients will be monitored under NHF or another sufficient therapy for the next 12 month followed by another mean overnight transcutaneous PCO2 level measure.

SECONDARY OUTCOMES:
quality of life with Saint Georges Respiratory Questionnaire (SGRQ) | after 4 weeks, 8 weeks and 12 month
  SGRQ is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.

OTHER OUTCOMES:
sleep quality | baseline, after 4 weeks, after 8 weeks, after 12 month
  sleep quality, measured by sleep efficiency, e.g. total sleep time vs sleep period time from PSG report.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Ambrock
Locations (1):
- Helios Klinik Ambrock, Hagen, North Rhine-Westphalia, Germany